CLINICAL TRIAL: NCT02505646
Title: Fluid Responsiveness Evaluation by AbdomiNal Compression in Kids Based on the STARLING Concept
Acronym: FRANCK
Status: Completed | Type: Observational
Sponsor: Hopital Louis Pradel (Other)
Responsible Party: Principal Investigator, Matthias Jacquet-Lagrèze, Dr Matthias Jacquet-Lagèze, Hopital Louis Pradel
Other Study IDs: EudraCT/ANSM 2015-A00388-41
Record Dates: First submitted 2015-07-16; First posted 2015-07-22 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Circulatory Failure
Keywords: circulatory failure; fluid responsiveness; abdominal compression
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observational study. No special intervention will be made — Data will be recorded in a context of fluid load in a context of circulatory failure. Stroke volume will be monitored, before, after an abdominal compression and after a fluid load.

SUMMARY:
Purpose:

Fluid responsiveness in a context of circulatory failure can be predicted by different way. Dynamic criteria such as pulse pressure variation, stroke volume variation during an end-expiratory occlusion maneuver or a passive leg raising have been reported to predict fluid responsiveness. Only aortic velocity peak variation measured with transthoracic echocardiography during mechanical ventilation has been reported to predict fluid responsiveness in children. Besides some physician use a maneuver of abdominal compression to predict fluid responsiveness in children with circulatory failure. This strategy has never been formally evaluated.

The investigators will study the diagnosis accuracy of the stroke volume variation induced by an abdominal compression to predict stroke volume variation after 10 ml/kg fluid load in children with circulatory failure.

Thirty-eight pediatric patients under eight years old in circulatory failure, for whom the attending physician has decided a fluid load will be included. Hemodynamic parameters: arterial pressure, heart rate, stroke volume measured with echocardiography; will be recorded. This data collection will be performed before, after abdominal compression and after a fluid load of 10 ml/kg.

Patients will be aposteriori sorted in two groups: Fluid responders and Fluid non-responders. Fluid responders are defined as patients that show an increase greater than 15 % in stroke volume. The diagnosis ability of the Stroke volume variation after an abdominal compression to predict fluid responsiveness will be investigate and receiving operative characteristic (ROC) curve will be built. The correlation between the variation of stroke volume during abdominal compression and during the fluid load will be studied. Other parameters such as arterial pressure and heart rate will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Age < 8 years old
* Patient with a circulatory failure defined as follow :

Treatment including vasopressor or inotrope

OR macrocirculatory failure

* Heart rate > 2 Standard Deviation (SD)
* Systolic arterial pressure < 2 SD
* Mean arterial pressure < 2 SD
* Diastolic arterial pressure < 2 SD

WITH signs of microcirculatory failure

* Capillary refill time > 2 secondes
* Blotch
* Organ dysfunction due to the circulatory failure (Oliguria < 0,5 ml/kg/h, acute lung injury, encephalopathy)

Exclusion Criteria:

* Opposition from the parents or the one who holds the parental authority
* Cardiogenic acute pulmonary edema,
* Extreme hemodynamic instability,
* Intra-abdominal hypertension,
* Recent abdominal surgery that does not permit an abdominal compression without causing pain.
* Patient with mechanical circulatory support, such as Extra Corporal Life Support or Berlin-Heart
* Patient with congenital cardiopathy with a palliative correction or an incomplete correction
* Open thorax
* Prone position
* Investigators not available
* No security number registration.
* Moribund patient

Max Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patient hospitalized in the intensive care unit of the hospital " feme mère enfant " or the cardiologic hospital of BRON who suffer from circulatory failure and for whom the attending physiscian has decided to administer a 10 ml/kg cristalloïd infusion.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Ability of the stroke volume variation after abdominal compression to predict fluid responsiveness | 30 minutes
  Stroke volume will be measured before and after a calibrated abdominal compression and after a fluid load. Patient will then be sorted in two groups. Responders defined as patient that show an increase in stroke volume after a 10ml/kg fluid load and Fluid non responders, defined as patient that show an increase of less than 15 % in stroke volume. The ROC curve will investigate the ability of stroke volume variation after abdominal compression to predict fluid responsiveness.

SECONDARY OUTCOMES:
Ability of the pulse pressure variation after abdominal compression to predict fluid responsiveness | 30 minutes
Ability of the heart rate variation after abdominal compression to predict fluid responsiveness | 30 minutes
Correlation between stroke volume variation, heart rate variation, pulse pressure variation between the abdominal compression and the fluid load | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Fellahi, MD, PhD, Study Director — Hôpital Louis Pradel, Hospice Civil de Lyon
Locations (2):
- France (2):
  - Intensive care and anesthesiology department, Hôpital Louis Pradel., Lyon
  - Pediatric Intensive care, Hôpital Femme Mère Enfant, Lyon

REFERENCES:
- [Derived] Jacquet-Lagreze M, Tiberghien N, Evain JN, Hanna N, Courtil-Teyssedre S, Lilot M, Baudin F, Chardonnal L, Bompard D, Koffel C, Portefaix A, Javouhey E, Fellahi JL. Diagnostic accuracy of a calibrated abdominal compression to predict fluid responsiveness in children. Br J Anaesth. 2018 Dec;121(6):1323-1331. doi: 10.1016/j.bja.2018.06.030. Epub 2018 Sep 6. PMID 30442260